CLINICAL TRIAL: NCT00676221
Title: Patient Reported Outcomes in Renal Transplant Patients Tolerating GI Symptoms Converted to Myfortic (EC-MPS).
Brief Title: Patient Reported Outcomes in Renal Transplant Patients Tolerating Gastrointestinal (GI) Symptoms Converted to Myfortic (EC-MPS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foothills Medical Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Serdar Yilmaz MD., PhD., FACS. Regional Chief, Div. of Transplant Surgery, Foothills Medical Centre, Div. of Transplant Surgery
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-20097
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Transplant
Keywords: Renal transplant recipient; Immunosuppression; Gastro-intestinal symptoms; Quality of life; Cellcept; Myfortic; Kidney transplant patients.
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Myfortic — Mycophenolate Mofetil (Cellcept) discontinued at Baseline visit. Mycophenolate Sodium(Myfortic)commenced the following day at equimolar doses orally BID.
  Cellcept 1000mg bid = Myfortic 720mg bid
  Other Names: EC-MPS

SUMMARY:
Hypothesis: Presently, some patients' mycophenolate mofetil (MMF.,Cellcept) related gastrointestinal (GI) symptoms are not being spontaneously reported. It is postulated that a conversion to enteric-coated mycophenolate sodium (EC-MPS.,Myfortic) from MMF will reduce the objectively measured GI symptom burden and improve GI-related quality of life.

Primary Objective: To determine the incidence of GI-related symptoms and the health related quality of life of renal transplant patients that are currently tolerating MMF. Assessed by GSRS and GIQLI.

Secondary Objective: To determine the impact on GI symptoms and the health related quality of life of renal transplant patients converted from MMF to Myfortic. Assessed by GSRS and GIQLI.

DETAILED DESCRIPTION:
Investigator originated proposal. Single centre-Foothills Medical Centre, Southern Alberta Transplant Program.

Study design: Three month, longitudinal, open-label, single arm study. Number of study visits: 3 (Baseline, 4-6 weeks, 12 weeks)

Planned sample size :Approx. 110 subjects. Study population will be primary or secondary renal transplant recipients who are stable and are on maintenance immunosuppressive medication which includes MMF.

Gastrointestinal rating scale (GSRS) and Gastrointestinal Quality of Life Index (GIQLI)will be the evaluation tool for GI symptoms, completed by study subject via a "touch screen" pc. at baseline, 4-6 week and final 12 week visit.

Study subjects will discontinue MMF following the evening dose on the day of Baseline visit and commence EC-MPS at equimolar doses of subject's current MMF dose.

At Final study visit (Week 12) study subject will be given the option of continuing on EC-MPS or resuming MMF.

Endpoints:

Primary: Incidence of patients tolerating MMF related GI symptoms.

Secondary:

1. Patient reported symptoms and quality of life after conversion from MMF to EC-MPS.
2. Adverse events.
3. Renal function as determined by Cockroft-Gault equation
4. Routine hematological and chemistry bloodwork.

Statistical consideration: Descriptive, pair T-Test analysis.

ELIGIBILITY:
Inclusion Criteria:

* Stable primary or secondary renal transplant recipients, males and females. 18-75 years of age.
* Stable GFR (>30ml/min) Cockroft-Gault equation at time of last clinic visit and at Screening/Baseline visit.
* Immunosuppression drug regimen that includes MMF(Cellcept)for at least 4 weeks prior to study enrollment.
* Renal transplant recipients who are tolerating or willing to tolerate GI symptoms related to MMF.
* Patients willing and capable of given written informed consent for study participation.

Exclusion Criteria:

* Non-stable renal transplant recipients ( infection, thrombocytopenia,neutropenia, anemia, fluctuating GFR, acute rejection < 1 week prior to study enrollment etc.)
* Malignancies other than treated basal cell and squamous cell carcinoma of the skin.
* Other serious medical conditions ( uncontrolled diabetes, peptic ulcers, etc)
* GI symptoms not related to MMF (ie infectious diarrhoea)
* Women of childbearing potential who are unwilling to use effective means of contraception.
* Presence of psychiatric illness that would interfere with study requ1rements.
* Ongoing acute medical intervention or hospitalization.
* Patients receiving any investigational drug or having received any investigational drug within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-08 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of GI related symptoms (GSRS) and the health related quality of life (GIQLI) of renal transplant recipients who are currently tolerating or willing to tolerate MMF. | 12 weeks

SECONDARY OUTCOMES:
To determine the impact on GI symptoms and the health related quality of life of renal transplant patients converted from MMF to EC-MPS. | 12 weeks
Adverse events. | 12 weeks
Renal function as determined by Cockroft-Gault equation. | 12 weeks
Routine hematological and biochemical bloodwork changes. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Yilmaz, MD., PhD, Principal Investigator — Foothills Medical Centre, Div. of Transplant Surgery
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada